CLINICAL TRIAL: NCT01605019
Title: A Multi-Center Clinical Pilot-Study to Evaluate the Performance of CoSeal in Reducing Post-Op Bleeding, Air Micro Emboli, and Cardiac Tissue Adhesions in Patients With Left Ventricular Assist Devices (LVADs)
Brief Title: The Use of CoSeal (Sealant Agent) in Patients During Left Ventricular Assist Device Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding for study stopped
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Brian A. Bruckner, M.D., Assistant Professor, Division of Cardiac & Transplant Surgery., The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00007027; BS11-000540 (Other: Baxter Healthcare Grant BS11-000540)
Record Dates: First submitted 2012-05-21; First posted 2012-05-24 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure; Ventricular Dysfunction
Keywords: Ventricular Assist Devices; Heart assist pumps; heart pumps; sealant agents
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CoSeal Arm (Experimental): patient randomized to received Coseal during LVAD implantation
  Interventions: Device: CoSeal
- BioGlue® Surgical Adhesive (Placebo Comparator): BioGlue® Surgical Adhesive or use of no sealant application
  Interventions: Device: BioGlue® Surgical Adhesive

INTERVENTIONS:
Device: CoSeal — 3 - 8mls of Coseal
  Arms: CoSeal Arm
Device: BioGlue® Surgical Adhesive — Total amount applied - 8 mls
  Other Names: Control - BioGlue® Surgical Adhesive or use of no sealant
  Arms: BioGlue® Surgical Adhesive

SUMMARY:
The purpose of this study is to evaluate the use of a device called CoSeal™. CoSeal™ is an FDA approved synthetic (man-made) surgical sealant which is currently used to help stop leaks in blood vessels during surgery.

This study is evaluating CoSeal™ when it is applied to various areas of the heart during the surgery to implant a Left Ventricular Assist Device (LVAD). the investigators are looking for evidence which indicates that CoSeal™ may be useful in reducing or stopping bleeding, the occurrence of micro emboli (small particles of air or blood), and the formation of cardiac adhesions (scar tissue strands that may form around the heart in the area of a previous LVAD operation) in patients who undergo LVAD implantation surgery.

DETAILED DESCRIPTION:
This is a prospective, single-blind (subjects and surgeon evaluator are blinded), randomized, multi-center, pilot study which is designed to evaluate the effects of CoSeal™ when used during a surgical procedure to implant a LVAD. The study sample size is 30 subjects; subjects will be randomized in a 2:1 fashion, 20 subjects will be randomized to CoSeal™ in the Treatment Group and 10 subjects will be randomized to no sealant in the Control Group. Bioglue will be used in the control group, only if necessary.

The Primary Objective of this prospective pilot study is to evaluate the use of CoSeal™ for its ability to reduce bleeding following the implantation of a LVAD. The secondary objectives will evaluate the use of CoSeal for its ability to reduce micro emboli during the LVAD implant procedure and prevent tissue adhesions following the implantation of a LVAD.

CoSeal™ (Baxter, Deerfield, Ill., USA) is a synthetic hydrogel consisting of two solutions of high molecular weight of polyethylene glycol which are co-extruded with a liquid sodium phosphate buffer from a syringe housing unit. The device is approved by the FDA for use in vascular reconstructions to achieve adjunctive hemostasis by mechanically sealing areas of leakage and it has been shown to provide superior anastomatic suture line sealing. In 2005, the CoSeal™ medical device was also approved in Europe and Australia for use in patients undergoing cardiac surgery to prevent or reduce the incidence, severity, and extent of post-surgical adhesions.

Data from this study will not be used to support any labeling changes. This is a PI initiative study that was submitted and granted funding from Baxter Healthcare for data and publishing of study data.

ELIGIBILITY:
Inclusion Criteria:

* Subject or the subject's legal representative has signed the IRB approved study informed consent.
* Subject is greater than or equal to 18 years of age.
* Subject has a known indication for implantation of a LVAD and meets the requirements for its implantation.
* Subject who, in the opinion of the investigator, will not require removal of the LVAD earlier than 6 weeks after implantation.

Exclusion Criteria:

* Subject requires the concomitant use of any other anti-adhesion product during LVAD implantation.
* Subject has an immune system disorder, immuno-deficiencies, or immuno-suppression.
* Subject has known hypersensitivity to the study device, CoSeal™, or any component of the study device.
* Subject is currently participating in another clinical trial for adhesion prevention or sealing evaluation and/or who has received such an investigational drug or device within the previous 30 days.
* Subject has previously undergone a LVAD implantation/explantation.
* Subject is pregnant or currently breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Bruckner, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (2):
- United States (2):
  - Texas Heart Institute, Houston, Texas
  - The Methodist Hospital DeBakey Heart & Vascular Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Data sharing plan to be determined.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CoSeal Arm | BioGlue® Surgical Adhesive
Started | 4 | 0
Completed | 1 | 0
Not Completed | 3 | 0
Not completed — pt did not meet transplant endpoint | 3 | 0

BASELINE CHARACTERISTICS:
Population: no data was analyzed - there were 4 subjects enrolled but the study was not completed due to discontinuation of funding therefore no data was analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | CoSeal Arm | BioGlue® Surgical Adhesive | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical — Data was collected for baseline and procedure but not outcome data was not collected on the 4 subjects that were enrolled prior to the study closure. Outcome data was not collected due to study discontinued due to lack of funding.
Sex: Female, Male — No baseline data collected because study was discontinued due to lack of funding

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduced Bleeding Following the Implantation of a LVAD
Description: The Primary Objective of this prospective pilot study is to evaluate the use of CoSeal™ for its ability to reduce bleeding following the implantation of a LVAD. Total output amounts for each chest tube (CT) will be collected every 24 hours until all chest tubes are discontinued. Additionally, the total number of blood transfusions required during the hospitalization to implant the LVAD will be collected
Time Frame: Participants will be follwed for the duration of hospital stay for LVAD implant, typically an average of 1-4 weeks.
Population: no analysis was performed on the 4 subjects enrolled in the study - they did not complete study.
Arm/Group | CoSeal Arm | BioGlue® Surgical Adhesive
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Evaluate the Use of CoSeal for Its Ability to Reduce Micro Emboli During the LVAD Implant Procedure and Prevent Tissue Adhesions Following the Implantation of a LVAD
Description: During the LVAD implant surgery, TEE and Transcranial Doppler will be conducted before and after the LVAD implant/CoSeal™ administration to detect possible micro emboli in the left ventricle (TEE) and in the intra-cranial circulation (TCD).
  • Intra-operative evaluation of surgical adhesions during LVAD explantation/heart transplant.
Time Frame: Participants will be followed for duration of hospital stay, typically average of 1-4 weeks at time of LVAD surgery & again at time of heart transplant surgery
Population: Analysis not completed - study terminated due to funding pulled by sponsor
Arm/Group | CoSeal Arm | BioGlue® Surgical Adhesive
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | CoSeal Arm | BioGlue® Surgical Adhesive
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

LIMITATIONS AND CAVEATS:
Only 4 subjects were enrolled in study prior to study being closed due to funding being pulled by grant sponsor.

Data was collected on their surgery and recovery but not analyzed due to limited sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less